CLINICAL TRIAL: NCT06695637
Title: Individualized Neuromodulation of Craving Control for Meth Use Disorders
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Key study staff left the university
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PSYCH-2023-32513
Record Dates: First submitted 2024-10-15; First posted 2024-11-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Substance Use Disorders; Methamphetamine Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Individuals diagnosed with MUDs randomized for study intervention
  Interventions: Radiation: active cTBS
- Sham control group (Sham Comparator): Individuals diagnosed with MUDs randomized for sham intervention
  Interventions: Radiation: sham cTBS

INTERVENTIONS:
Radiation: active cTBS — Transcranial Magnetic Stimulation (TMS) is a non-invasive neuromodulation technique which employs magnetic fields to stimulate neural activity in the brain. cTBS is a specific TMS protocol, wherein bursts of high-frequency magnetic pulses are repeatedly applied in a rhythmic pattern, mimicking the theta rhythm of neural oscillations. Studies suggest that cTBS has the potential to modulate cortical excitability and synaptic plasticity, leading to alterations in targeted brain function.
  Baseline measures will be collected to develop individualized targets for stimulation and also understand how brain structure and activity may change in response to cTBS.
  Arms: Study group
Radiation: sham cTBS — The intervention group receives cTBS and the control group receives sham stimulation using the sham option in the coil that makes the same noise and feeling without delivering significant amount of magnetic energy into the brain. Both groups are exposed to drug and neutral pictures before and after receiving stimulation. People in the active group will receive cTBS with corrected individualized stimulation intensity to have 1 V/m in targeted brain regions while in the sham group people will only receive sham condition with a similar look, sound, and feel of active stimulation.
  Arms: Sham control group

SUMMARY:
Drug craving is one of the key aspects of substance use disorders (SUDs) and is associated with continued drug use and relapse. Approximately 70% of those entering treatment will relapse within one year. To improve treatment outcomes, new interventions targeting the underlying brain biomarkers of relapse vulnerability hold significant promise in reducing this critical public health problem.

This clinical trial is designed as a randomized, double-blind, sham-controlled study, aiming to investigate the effects of continuous theta burst stimulation (cTBS) on individuals diagnosed with Methamphetamine Use Disorders (MUDs). Only adults (22-65 years old) who are already living in an abstinence-based residential setting for substance use treatment will be recruited, and participants will be escorted to and from the MIDB center for their imaging and brain stimulation sessions. After a baseline assessment to determine eligibility, the study will include 40 participants, who will be randomly assigned to two groups: the active cTBS group and the sham cTBS group (a control group receiving a placebo treatment).

ELIGIBILITY:
Inclusion Criteria:

* Abstinent from any substance or alcohol use (excluding caffeine or nicotine) for a minimum of 1 week at study enrollment
* Has the intention to remain in their treatment program(s) until the end of the intervention portion of the study.
* Able to provide written consent and comply with study procedures.
* Meets the DSM-V MINI diagnostic criteria for methamphetamine use disorder (MUD).
* Subjects may have current comorbid drug use, but one of their major substance use disorder diagnosis needs to be methamphetamine use. Potential subjects will not be excluded for being on medication-assisted treatments (MATs), such as those used to treat substance use disorders.

Exclusion Criteria:

* Any contraindications for MRI scanning (up to the discretion of MIDB staff:

metal implants, pacemakers or any other implanted electrical device, injury with metal, braces, dental implants, non-removable body piercings, pregnancy, breathing or moving disorder, moderate to severe heart disease).

* Any medical condition or treatment with neurological sequelae (i.e., stroke, tumor, HIV, intracranial lesions)
* Having epilepsy, a personal history of a seizure (beyond fever or withdrawal or medical induced seizure), or individuals with a family history of clinically proven epilepsy disorder in a first degree relative
* Over 9 months of abstinence from substance use
* A head injury resulting in a loss of consciousness exceeding 30 minutes (i.e., moderate or severe TBI)
* Presence of a condition that would render study measures difficult or impossible to administer or interpret
* Age outside the range of 22 to 65
* Entrance to the treatment program under a court mandate. (i.e., legally incarcerated)
* History of ECT or cortical energy exposure within the past 6 months, including participation in any other neuromodulation studies
* Being pregnant. For females of reproductive potential: negative pregnancy test or use of highly effective contraception for at least 1 month prior to baseline will be necessary for inclusion.
* Having current active suicidal ideations reported in baseline psychiatry interview
* Having active bipolar disorder (with a risk of mania)
* Using medications that significantly increase risk of seizure for this study based on the clinical judgement of the study's medical team such as immediate release bupropion (Wellbutrin IR), stimulants, and tramadol.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Connectivity between the Amygdala/Ventral Striatum and Frontopolar Cortex Measurement | baseline, 24 hours
  Connectivity strength between the amygdala/ventral striatum and frontopolar cortex, measured by generalized psychophysiological interaction (gPPI) analysis.
  Measurement Tool: Connectivity strength measured using fMRI-based gPPI with Brainnetome atlas parcellation.
  Unit of Measure: Regression coefficient representing connectivity strength.

SECONDARY OUTCOMES:
Change in Self-Reported Craving in Methamphetamine Use Disorder (MUD) | baseline, 24 hours
  Self-reported craving levels in response to continuous theta-burst stimulation (cTBS).
  Measurement Tool: Craving levels assessed via a standardized self-report craving scale (e.g., Visual Analog Scale for Craving or other validated scale for substance use disorders).
  Unit of Measure: Score change or percentage change from baseline on the craving scale.
Baseline Connectivity Predicting Neural and Subjective Response to Individualized cTBS | baseline, 24hours
  Baseline connectivity between the amygdala/ventral striatum and frontopolar cortex as a predictor of neural and subjective response to individualized cTBS.
  Measurement Tool: Baseline connectivity measured using fMRI-based generalized psychophysiological interaction (gPPI) analysis with Brainnetome atlas parcellation; response measured by self-report craving scale and fMRI post-intervention.
  Unit of Measure: Predictive accuracy for post-intervention craving scores (score change or percentage change) and neural activity (correlation coefficients).
Predictive Role of Individualized Current Density in Prefrontal Cortex for Subjective and Neural Response to cTBS density in the head models in the prefrontal cortex in both subjective and neural response to cTBS | baseline, 24 hours
  Outcome Measure Title/Description: Current density within the prefrontal cortex, estimated from individualized head models, as a predictor of subjective craving response and neural response following cTBS.
  Measurement Tool: Current density calculated from structural MRI-based individualized head models, with predictive accuracy assessed through self-report craving scale scores and fMRI measures post-intervention.
  Unit of Measure: Current density (A/m²) for neural prediction; craving response measured by score or percentage change on craving scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lim, MD, Principal Investigator — University of Minnesota